CLINICAL TRIAL: NCT03748212
Title: A Randomized, Open-label, Fed, Single Dose, Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-385 in Healthy Volunteers
Brief Title: Clinical Trial to Evaluate Pharmacokinetic Profiles and Safety Between CKD-385 and D935 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 188BE18024
Record Dates: First submitted 2018-11-18; First posted 2018-11-20 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Hypertension
Keywords: Hypertension; Chronic stable angina; Congestive Heart Failure
MeSH Terms: conditions — Hypertension; Angina, Stable; Heart Failure | interventions — D 935

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): D935 Cap. 1T
  Interventions: Drug: D935 Cap. 1T
- Group 2 (Experimental): CKD-385 Tab. 1T
  Interventions: Drug: CKD-385 Tab. 1T

INTERVENTIONS:
Drug: D935 Cap. 1T — single oral administration under fed condition
  Other Names: D935
  Arms: Group 1
Drug: CKD-385 Tab. 1T — single oral administration under fed condition
  Other Names: CKD-385
  Arms: Group 2

SUMMARY:
A randomized, open-label, fed, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-385 in healthy volunteers

DETAILED DESCRIPTION:
To healthy subjects of 52, following treatments are administered dosing in each period and wash-out period is a minimum of 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy adult aged over 19 at the time of screening
2. Weight over 55, with BMI between 17.5kg/m² and 30.5kg/m²
3. Subject who has no congenital or chronic disease within the last 3 years and no medical symptoms or signs as a result of medical examination
4. Suitable subject who is determined at the time of screening by examiners according to the characteristics of the medicine such as hematology test, blood chemistry test, urine test, virus / bacteriological test, vital signs, electrocardiogram test
5. Subject who signed the written consent form approved by Chonbuk National University Hospital IRB to participate in this study with full understanding of the purpose and contents of the examination prior to participation of the clinical trial
6. Subject who has the ability and willingness to participate in the clinical trial

Exclusion Criteria:

1. Subject who has (or has histories of) clinically significant blood, kidney, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, liver, mental, neurological or allergic diseases(except for asymptomatic seasonal allergy at the time of administration) or evidence(except for simple dental history such as dental calculus, impacted tooth, wisdom tooth, etc.)
2. Subject with a history of gastrointestinal disorders(esophageal achalasia or esophagus stenosis, Crohn's disease) or gastrointestinal surgery(except for simple appendicitis surgery or hernia surgery or tooth extraction surgery) that may affect the absorption of drug
3. Subject who shows the following values as a result of laboratory tests

   *ALT or AST > 2 times upper limit of normal range
4. Subject who has a history of regular alcohol consumption in excess of 210 g/week within 6 months of screening
5. Subject who smokes more than one pack of cigarette a day within 6 months of screening
6. Subject who took other clinical trial drugs or bioequivalence test drugs within 3 months before the first administration of clinical trial drug
7. Subject who conform to the specific items below

   * systolic blood pressure less than 90 mmHg, greater than 140 mmHg or diastolic blood pressure less than 60 mmHg or greater than 90 mmHg in a sitting position
   * Severe bradycardia (less than 50 beats/minute)
8. Subject who has significant alcohol abuse or drug abuse within a year of screening
9. Subject who took drugs which are known as disturbing drug metabolism within 30 days prior to the first administration of clinical trial drug.
10. Subject who uses any of other drugs, including over-the-counter medications and prescription medications within 10 days prior to first administration of clinical trial drug.
11. Subject who donated whole blood within 2 months prior to first administration of clinical trial drug or blood components within 1 month prior to first administration of clinical trial drug
12. Subject who is hypersensitive to the components of a clinical trial drug or clinical trial drug itself.
13. Subject who does not consent to reliable contraception during the entire period of clinical trial and until 7th day of administration of clinical trial drug.
14. Subject who is not able to consume high-fat meal provided during the clinical trial
15. Any other subject who is decided by investigators to be ineligible in clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-10-24 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
AUCt of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Area under the plasma concentration of Carvedilol verses time curve from time zero to time of last quantifiable concentration
Cmax of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Maximum plasma concentration of Carvedilol

SECONDARY OUTCOMES:
AUCinf of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Area under the plasma concentration of Carvedilol versus time curve from time zero to time infinity
Tmax of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Time to maximum concentration of Carvedilol
t1/2 of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Terminal elimination half-life of Carvedilol
CL/F of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Total body clearance of Carvedilol
Vd/F of Carvedilol | Pre-dose(0hr), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48hrs
  Apparent volume of distribution of Carvedilol

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Ho Jang, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No